CLINICAL TRIAL: NCT02347995
Title: Resistive Training Combined With Nutritional Therapy After Stroke
Acronym: REPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N1461-R; HP-00062067 (Other: Baltimore VAMC)
Record Dates: First submitted 2015-01-08; First posted 2015-01-28 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Exercise; Protein; Nutrition; Stroke
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistive Training (Placebo Comparator): Participants will drink a placebo beverage after each resistance training session.
  Interventions: Other: Placebo
- Resistive Training + Protein (Experimental): Participants will drink 30 grams of whey protein after each resistance training session.
  Interventions: Other: Protein

INTERVENTIONS:
Other: Protein — This training is designed to target the major muscle groups of the leg. Resistance training will be completed through a combination of lower extremity machines and complemented by whole body exercises such as squatting. The lower extremity machines include leg press, leg extension, and leg curl. This group will drink a beverage containing protein after each training session.
  Arms: Resistive Training + Protein
Other: Placebo — This training is designed to target the major muscle groups of the leg. Resistance training will be completed through a combination of lower extremity machines and complemented by whole body exercises such as squatting. The lower extremity machines include leg press, leg extension, and leg curl.This group will drink a placebo beverage after each training session.
  Arms: Resistive Training

SUMMARY:
Stroke survivors experience severe muscle wasting during the chronic phase of recovery, with implications for strength, function and general health. Although resistive exercise training effectively combats this problem, it is unknown whether sub-optimal protein intake limits the observed gains in skeletal muscle growth. Skeletal muscle adaptations may occur when resistive training (RT) is combined with nutritional therapy in the form of post- exercise protein consumption. This study would be the first to directly compare RT+protein supplementation to RT+placebo (same calories as protein supplement) in those with chronic hemiparesis caused by stroke, providing evidence-based rationale for combination therapy in the clinical care of this population.

DETAILED DESCRIPTION:
The VA research team has played a prominent role in documenting the significant skeletal muscle atrophy that accompanies chronic hemiparesis after disabling stroke. Muscle volume is reduced by 24% in paretic vs. non-paretic legs, having significant implications for strength, function, fitness, metabolism and general health. The investigators' previous work establishes progressive, high-intensity resistive training (RT) as an effective rehabilitation strategy for older stroke survivors, producing thigh muscle hypertrophy on both the paretic and non-paretic sides. Protein supplementation can significantly augment gains in muscle mass after RT in healthy populations, but no experiments have yet been conducted in stroke. New preliminary data from the investigators' group indicates that stroke participants consume 20% less protein than the recommended daily amount for older individuals (0.80 vs. 1.0 g/kg/day) suggesting that relative gains in skeletal muscle could be significantly better in the presence of adequate protein intake. New data also indicates that leg muscle mass predicts resting metabolic rate (RMR) in stroke, implying that a combined nutrition and RT therapy aimed at maximizing muscle gains would translate into improved energy balance, a key factor in rehabilitation success. A better understanding of the true potential for aggressive RT interventions to address stroke-related atrophy and related problems for maximum benefit awaits clinical trials directly comparing RT with and without nutritional therapy. The investigators propose to conduct a 12-week randomized placebo controlled clinical trial comparing the effects of RT+ protein supplementation at 1.2 g/kg/day (RT+PRO) vs. RT+isocaloric placebo (RT+PLA) on body composition, hypertrophy, strength, functional mobility and energy expenditure in chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Stroke > 3 months prior
* Completion of all regular post-stroke physical therapy
* Adequate language and neurocognitive function to participate in testing and training and to provide informed consent
* Able to walk 10 meters without human assistance

Exclusion Criteria:

* Regular structured resistive exercise (>2x/week)
* Alcohol consumption >3oz. liquor, 3 x 4oz. glasses of wine, or 3 x 12oz beers/day, by self report
* Neurological history of: a) dementia by clinical evaluation, b) severe receptive or global aphasia, which confounds testing and training, operationally defined as unable to follow 2 point commands, c) untreated major depression by clinical interview
* Medical History: a) recent hospitalization (less than 3 months prior to study entry) for severe medical disease, b) orthopedic or chronic pain condition restricting exercise, c) pulmonary or renal failure, d) active cancer, e) untreated poorly controlled hypertension measured on at least 2 occasions (greater than 190/100) f) untreated and / or poorly controlled diabetes with fasting blood glucose of greater than 170 and HbA1c greater than 10.0, g) medications: oral steroids, h) currently pregnant
* Cardiac history of: a) unstable angina, b) recent (less than 3 months prior to study entry) myocardial infarction, congestive heart failure (NYHA category II-IV); c) hemodynamically significant valvular dysfunction
* Any medical condition that, in the opinion of the Investigator, might interfere with the subject's participation in the study, poses any added risk for the subject, or confounds the assessment of the subject

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in thigh muscle area | Measured at baseline and after the 3 month intervention
  muscle area in cm2

SECONDARY OUTCOMES:
Change in muscle strength | Measured at baseline and after the 3 month intervention
  strength
Change in functional mobility (6 min walk distance) | Measured at baseline and after the 3 month intervention
  6 min walk distance
Change in myostatin messenger RNA (mRNA) level | Measured at baseline and after the 3 month intervention
  myostatin mRNA (AU)

CONTACTS AND LOCATIONS:
Overall Officials: Alice S. Ryan, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryan AS, Novitskaya M, Treuth AL. Predictive Equations Overestimate Resting Metabolic Rate in Survivors of Chronic Stroke. Arch Phys Med Rehabil. 2022 Jul;103(7):1352-1359. doi: 10.1016/j.apmr.2022.01.155. Epub 2022 Feb 19. PMID 35192798